CLINICAL TRIAL: NCT07191067
Title: A Multi-Center Two-Arm, Randomized, Blinded, Sham-Controlled Trial to Determine the Safety and Efficacy of the NOVABLOC System on Postoperative Pain, Functional Recovery and Opioid Use in Patients Undergoing Primary Total Knee Arthroplasty
Brief Title: Pivotal Study on the NOVABLOC System for Patients Undergoing Primary Total Knee Arthroplasty
Acronym: NOVABLOC TKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Synaptrix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1-25-001
Record Dates: First submitted 2025-09-08; First posted 2025-09-24 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- NOVABLOC Stimulation (Active Comparator): Subjects will receive NOVABLOC stimulation prior to their TKA
  Interventions: Device: Percutaneous radiofrequency electrical nerve stimulation
- Sham Stimulation (Sham Comparator): Subject will receive sham non-therapeutic stimulation
  Interventions: Device: Non-therapeutic stimulation

INTERVENTIONS:
Device: Percutaneous radiofrequency electrical nerve stimulation — Percutaneous radiofrequency electrical nerve stimulation will be applied to the femoral and sciatic nerves prior to TKA.
  Arms: NOVABLOC Stimulation
Device: Non-therapeutic stimulation — Electrical square wave stimulation performed to mimic the duration of the active arm and mimic the procedure for blinding purposes.
  Arms: Sham Stimulation

SUMMARY:
Multi-center, randomized, blinded, sham-controlled study to determin the safety and efficacy of the NOVABLOC system on post-operative pain in patients undergoing TKA procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant females age ≥ 21 years of age;
2. Has an underlying diagnosis of osteoarthritis indicated for a primary unilateral TKA according to established treatment guidelines;
3. Able and willing to provide and document informed consent and Authorization for Release of Protected Health Information (PHI);
4. Able and willing to comply with all trial tests, procedures, assessments, and follow-up visits for up to 45 days.
5. Able to read and understand instructions and information presented in English.

Exclusion Criteria:

1. Chronic opioid use (average ≥ 30 oral morphine equivalents / day) ≤ thirty (30) days of the TKA procedure;
2. Extended-release or long-acting opioid (e.g. buprenorphine, Morphine ER, etc.) use ≤ thirty (30) days of the TKA procedure;
3. History of substance abuse or misuse;
4. History of significant cardiac disease (e.g. ejection fraction ≤ 50%; coronary intervention ≤ six (6) months; significant valvular abnormalities);
5. Prior radiofrequency ablation or cryotherapy for pain on the operative knee;
6. Prior TKA on the operative knee;
7. BMI > 40;
8. History of neurological, neuromuscular or neuropathic disease that would confound the study results, including chronic pain conditions;
9. Have an active implanted biomedical device (such as cardiac pacemaker, insulin pump, pain stimulator, implantable cardioverter defibrillator) or cochlear [ear] stimulator);
10. History of hip or knee dislocation or bone fractures on the operative leg;
11. Sepsis or systemic infectious illness; local infection of skin or subcutaneous tissues where procedural access is required including thigh, hip or groin;
12. Concomitant medical or psychiatric illness that could compromise evaluation or treatment, including anxiety (GAD-7 score >10) or depression (PHQ-9 score >15);
13. Pregnant, actively planning a pregnancy or breast-feeding a child;
14. Uncontrolled diabetes (A1C > 7.5%);
15. History of bleeding disorder;
16. Participating in another clinical trial/investigation within 45 days prior to signing informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Worst Pain at Day 10 | 10 days post-TKA
  The worst pain felt by each subject at day 10 after the TKA procedure (as measured by question 3 on the BPI)

SECONDARY OUTCOMES:
Total morphine equivalents used | 5 days post-TKA
  Total morphine equivalents used cumulatively through Day 5

CONTACTS AND LOCATIONS:
Locations (1):
- Alabama Orthopedic Sports Medicine & Baldwin County Surgery Center, Daphne, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided